CLINICAL TRIAL: NCT07005895
Title: Feasibility of Using the Gatorade Sports Science Institute (GSSI) Labs App for Hydration Related Outcomes: User Engagement and Individual Variability of Transdermal Optical Imaging Features Before and After Acute Fluid Ingestion
Brief Title: Feasibility of Using the Gatorade Sports Science Institute (GSSI) Labs App for Hydration Related Outcomes
Status: Recruiting | Type: Observational
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-2503
Record Dates: First submitted 2025-05-12; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Hydration
Keywords: transdermal optical imaging; TOI; app; user engagement
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adult user of a wearable activity tracker: Male or female 18-65 who wears their own activity tracker daily
  Interventions: Other: Hydration assessment via mobile app

INTERVENTIONS:
Other: Hydration assessment via mobile app — Open the Gatorade Sports Science Institute (GSSI) branded mobile application and click on 'Complete Hydration Assessment'

SUMMARY:
This remote study will evaluate the feasibility of using the Gatorade Sports Science Institute (GSSI) Labs App for remotely collecting hydration related outcomes.

DETAILED DESCRIPTION:
The primary objective is to understand user engagement and feasibility of remotely collecting subjective and self-reported markers of hydration status as well as markers of hydration using transdermal optical imaging (TOI) within the Gatorade Sports Science Institute (GSSI) branded mobile application (adherence and dropout rates, and differences between demographics). The secondary objective is to understand the within subject variability of TOI features before and after acute fluid ingestion during remote data collection.

Tertiary objectives are to compare self-reported measures of hydration status against the TOI hydration model prediction before and after acute fluid ingestion during remote data collection.

An outside service was contracted for recruiting. Please do not contact the investigator to express interest.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age, inclusive
* Male or female. If female, subject is not pregnant, planning to get pregnant, or currently breast feeding
* Able to speak, write, and read English
* Provision of written consent to participate
* Owns and wears an activity tracker daily, including during sleep, except when submerged underwater (i.e., swimming, bathing) and is willing to connect their device to the app, per GSSI Labs App requirements (Oura, WHOOP, Apple Watch, Garmin, Polar, Withings, or Fitbit).
* Owns a bathroom scale
* Able to drink 600mL (600 mL = 20 oz = 2 ½ cups) of water as directed.
* Willing to avoid alcohol consumption 24 hours prior to study session(s)

Exclusion Criteria:

* Subject is currently enrolled in a clinical trial or has participated in a clinical trial within the past 30 days.
* Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If subject is unsure if a company would be considered a competitor to Gatorade, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Activity tracker-wearing adult
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
User engagement and feasibility: Subjective and self-reported markers of hydration status | At two identical 2-hour study sessions with at least one full day and a maximum of 6 days in between study sessions
  Understand user engagement and feasibility of remotely collecting subjective and self-reported markers of hydration status
User engagement and feasibility: Markers of hydration using transdermal optical imaging (TOI) | At two identical 2-hour study sessions with at least one full day and a maximum of 6 days in between study sessions
  Understand user engagement and feasibility of remotely collecting markers of hydration using transdermal optical imaging (TOI)

SECONDARY OUTCOMES:
Understand the within subject variability of TOI features before and after acute fluid ingestion during remote data collection | At two identical 2-hour study sessions with at least one full day and a maximum of 6 days in between study sessions
  Within subject variation in the tertiary outcomes listed in Other Pre-specified Outcomes 4-7

OTHER OUTCOMES:
Self-reported measure of hydration status: Body mass | Before and after acute fluid ingestion during remote data collection at two identical 2-hour study sessions with at least one full day and a maximum of 6 days in between study sessions
  Home scale body mass, against the TOI hydration model prediction
Self-reported measure of hydration status: Urine color | Before and after acute fluid ingestion during remote data collection at two identical 2-hour study sessions with at least one full day and a maximum of 6 days in between study sessions
  Urine color against the TOI hydration model prediction rated from very pale yellow to brown on a 7-color chart, against the TOI hydration model prediction
Self-reported measure of hydration status: Perceived thirst | Before and after acute fluid ingestion during remote data collection at two identical 2-hour study sessions with at least one full day and a maximum of 6 days in between study sessions
  Thirst rating in the app using a 7-point categorical scale, against the TOI hydration model prediction
Self-reported measure of hydration status: Feeling hydrated | Before and after acute fluid ingestion during remote data collection at two identical 2-hour study sessions with at least one full day and a maximum of 6 days in between study sessions
  Within the app, select Yes or No as to whether feeling sufficiently hydrated or not, against the TOI hydration model prediction

CONTACTS AND LOCATIONS:
Overall Officials: Shellen Goltz, PhD, RD, Principal Investigator — Advanced Personalized Ideation Center (API) & Gatorade Sports Science Institute (GSSI), PepsiCo Global R&D - Life Sciences
Locations (1):
- Advanced Personalized Ideation Center (API) and Gatorade Sports Science Institute (GSSI), PepsiCo Global R&D - Life Sciences, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No